CLINICAL TRIAL: NCT00849004
Title: Comparison of the Effectiveness in Prevention of Hypertrophic Scars or Keloids Between Silicone Sheet, Silicone Gel and Paper Steri-strip-A Randomised Controlled Trial.
Brief Title: Prevention of Hypertrophic Scars or Keloids
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Kuei-Chang Hsu, Consultant Surgeon, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 97CT1018; 97CT1018
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Hypertrophic Scars
Keywords: keloid; silicone sheet; silicone gel; paper tape; steri-strip
MeSH Terms: conditions — Cicatrix, Hypertrophic; Keloid | interventions — Silicone Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gel vs. Sheet (Active Comparator): One group will act to compare the effectiveness between silicone gel and silicone sheet.
  Interventions: Other: silicone gel; Other: silicone sheet
- sheet vs. paper tape (Active Comparator): The second group between silicone sheet and paper tape.
  Interventions: Other: silicone sheet; Other: paper tape
- gel vs. paper tape (Active Comparator): One group will act to compare the effectiveness between silicone gel and paper tape.
  Interventions: Other: silicone gel; Other: paper tape

INTERVENTIONS:
Other: silicone gel — silicone gel
  Arms: Gel vs. Sheet; gel vs. paper tape
Other: silicone sheet — silicone sheet
  Arms: Gel vs. Sheet; sheet vs. paper tape
Other: paper tape — paper tape
  Arms: gel vs. paper tape; sheet vs. paper tape

SUMMARY:
Keloids and hypertrophic scars are not major illness. However, their effects can be from causing pain and itch which substantially interfere daily activity to as severe as causing deformity and other functional impairment. For standard surgical wounds, taking median sternotomy wounds from open heart surgery and lower abdominal wounds from gynecological wounds for example, the incidence of these problems can be from 10% to 60%. To prevent or treat these problems, physicians have used many modalities. One of the most convenient, most cost-effective and most non-invasive methods for patients is using dressings like silicone sheets, silicone gels or paper tapes, which is on the list of 1st line choices of an international recommendation. According to a literature review, most of the previous studies on similar topics are either of small sample size, on non-standard wounds or comparisons between wounds on different patient groups. The methodologies of previous studies are thus not vigorous enough. To get the highest level of evidence on selecting the best dressings for preventing and treating keloids and hypertrophic scars, we will recruit about 75 patients and apply two selected dressings on each halves of their standard surgical wounds to compare their differences. The investigators hope the result of this study can help us find the best modality to use and can contribute to the welfare of our future patients.

DETAILED DESCRIPTION:
Patients who undergo gynecological surgery with transverse lower abdominal wounds and who undergo cardiovascular surgery with median sternotomy wounds in our hospital will be assessed. Those who have or will have diabetes, chemotherapy, radiotherapy and known history of allergy to silicone will be excluded. Altogether, about 75 patients will be recruited. Each patient's wound will be divided into two halves. One test dressing will be applied to a half, which is determined by random, and a different test dressing to the other half. The total 75 patients will thus be divided into 3 groups of 25 patients. One group will act to compare the effectiveness between silicone gel and silicone sheet, the second group between silicone sheet and paper tape, and the third group between silicone gel and paper tape. The dressings will be applied one week after surgery and at least 12 hours per day until 3 months after surgery. All patients will be followed up at 4 weeks, 8 weeks, 12 weeks, 6 months and 12 months. Three domains of outcomes will be measured. One is the appearance of the scars which will be rated with Vancouver scale, which has been proved to be a reliable scale.34 35 When rating with the Vancouver scale, standardised photographs of the scars will be taken in a standardised photo studio using a single high-resolution digital camera in a standardised light condition and at a fixed distance because any difference in photographic conditions will make difference in the Vancouver scores. The other two domains are pain and itching of the scars, which will be evaluated with Visual Analog Ratings (VAR). Pain and itching are very subjective, so the rating method should be very easy to understand and applicable for our patients and that is why we chose VAR as a tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo gynecological surgery with transverse lower abdominal wounds.
* Patients who undergo cardiovascular surgery with median sternotomy wounds in our hospital will be assessed.

Exclusion Criteria:

* Those who have or will have:

  * diabetes
  * chemotherapy
  * radiotherapy
* known history of allergy to silicone will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Scar appearance measured with Vancouver Scar Scores. | 12 months

SECONDARY OUTCOMES:
pain and itchiness measured with Visual Analog Scales. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Chang Hsu, surgeon, Principal Investigator — Department of plastic surgery in Kaohsiung Veterans General Hospital in Taiwan
Locations (1):
- Kaohsiung Veterans General Hospital: R.O.C., Kaohsiung City, Taiwan

REFERENCES:
- [Background] Pellard S. Epidemiology, aetiology and management of abnormal scarring: a review of the literature. J Wound Care. 2006 Jan;15(1):44-8. doi: 10.12968/jowc.2006.15.1.26863. PMID 16669306
- [Background] Murison M, James W. Preliminary evaluation of the efficacy of dermatix silicone gel in the reduction of scar elevation and pigmentation. J Plast Reconstr Aesthet Surg. 2006;59(4):437-9. doi: 10.1016/j.bjps.2005.09.037. No abstract available. PMID 16756266
- [Background] Rayner K. The use of pressure therapy to treat hypertrophic scarring. J Wound Care. 2000 Mar;9(3):151-3. No abstract available. PMID 11933297
- [Background] Mustoe TA. Scars and keloids. BMJ. 2004 Jun 5;328(7452):1329-30. doi: 10.1136/bmj.328.7452.1329. No abstract available. PMID 15178589
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427
- [Result] Wu WS, Wang FS, Yang KD, Huang CC, Kuo YR. Dexamethasone induction of keloid regression through effective suppression of VEGF expression and keloid fibroblast proliferation. J Invest Dermatol. 2006 Jun;126(6):1264-71. doi: 10.1038/sj.jid.5700274. PMID 16575391
- [Result] Giovannini UM. Treatment of scars by steroid injections. Wound Repair Regen. 2002 Mar-Apr;10(2):116-7. doi: 10.1046/j.1524-475x.2002.00206.x. No abstract available. PMID 12028527
- [Result] Chuangsuwanich A, Osathalert V, Muangsombut S. Self-adhesive silicone gel sheet: a treatment for hypertrophic scars and keloids. J Med Assoc Thai. 2000 Apr;83(4):439-44. PMID 10808705
- [Result] Suetak T, Sasai S, Zhen YX, Tagami H. Effects of silicone gel sheet on the stratum corneum hydration. Br J Plast Surg. 2000 Sep;53(6):503-7. doi: 10.1054/bjps.2000.3388. PMID 10927682
- [Result] Borgognoni L. Biological effects of silicone gel sheeting. Wound Repair Regen. 2002 Mar-Apr;10(2):118-21. doi: 10.1046/j.1524-475x.2002.00205.x. No abstract available. PMID 12028528
- [Result] Musgrave MA, Umraw N, Fish JS, Gomez M, Cartotto RC. The effect of silicone gel sheets on perfusion of hypertrophic burn scars. J Burn Care Rehabil. 2002 May-Jun;23(3):208-14. doi: 10.1097/00004630-200205000-00010. PMID 12032371
- [Result] Quinn KJ. Silicone gel in scar treatment. Burns Incl Therm Inj. 1987 Oct;13 Suppl:S33-40. doi: 10.1016/0305-4179(87)90091-x. No abstract available. PMID 3690373
- [Result] Ahn ST, Monafo WW, Mustoe TA. Topical silicone gel for the prevention and treatment of hypertrophic scar. Arch Surg. 1991 Apr;126(4):499-504. doi: 10.1001/archsurg.1991.01410280103016. PMID 2009067
- [Result] Katz BE. Silicone gel sheeting in scar therapy. Cutis. 1995 Jul;56(1):65-7. PMID 7555106
- [Result] Niessen FB, Spauwen PH, Robinson PH, Fidler V, Kon M. The use of silicone occlusive sheeting (Sil-K) and silicone occlusive gel (Epiderm) in the prevention of hypertrophic scar formation. Plast Reconstr Surg. 1998 Nov;102(6):1962-72. doi: 10.1097/00006534-199811000-00023. PMID 9810992
- [Result] Chan KY, Lau CL, Adeeb SM, Somasundaram S, Nasir-Zahari M. A randomized, placebo-controlled, double-blind, prospective clinical trial of silicone gel in prevention of hypertrophic scar development in median sternotomy wound. Plast Reconstr Surg. 2005 Sep 15;116(4):1013-20; discussion 1021-2. doi: 10.1097/01.prs.0000178397.05852.ce. PMID 16163087
- [Result] Atkinson JA, McKenna KT, Barnett AG, McGrath DJ, Rudd M. A randomized, controlled trial to determine the efficacy of paper tape in preventing hypertrophic scar formation in surgical incisions that traverse Langer's skin tension lines. Plast Reconstr Surg. 2005 Nov;116(6):1648-56; discussion 1657-8. doi: 10.1097/01.prs.0000187147.73963.a5. PMID 16267427
- [Result] Abergel RP, Dwyer RM, Meeker CA, Lask G, Kelly AP, Uitto J. Laser treatment of keloids: a clinical trial and an in vitro study with Nd:YAG laser. Lasers Surg Med. 1984;4(3):291-5. doi: 10.1002/lsm.1900040310. PMID 6390045
- [Result] Bouzari N, Davis SC, Nouri K. Laser treatment of keloids and hypertrophic scars. Int J Dermatol. 2007 Jan;46(1):80-8. doi: 10.1111/j.1365-4632.2007.03104.x. PMID 17214728
- [Result] Chan HH, Wong DS, Ho WS, Lam LK, Wei W. The use of pulsed dye laser for the prevention and treatment of hypertrophic scars in chinese persons. Dermatol Surg. 2004 Jul;30(7):987-94; discussion 994. doi: 10.1111/j.1524-4725.2004.30303.x. PMID 15209788
- [Result] McCraw JB, McCraw JA, McMellin A, Bettencourt N. Prevention of unfavorable scars using early pulse dye laser treatments: a preliminary report. Ann Plast Surg. 1999 Jan;42(1):7-14. doi: 10.1097/00000637-199901000-00002. PMID 9972711
- [Result] Kelly AP. Medical and surgical therapies for keloids. Dermatol Ther. 2004;17(2):212-8. doi: 10.1111/j.1396-0296.2004.04022.x. PMID 15113289
- [Result] Staley MJ, Richard RL. Use of pressure to treat hypertrophic burn scars. Adv Wound Care. 1997 May-Jun;10(3):44-6. PMID 9306778
- [Result] Macintyre L, Baird M. Pressure garments for use in the treatment of hypertrophic scars--a review of the problems associated with their use. Burns. 2006 Feb;32(1):10-5. doi: 10.1016/j.burns.2004.06.018. PMID 16413399
- [Result] Puzey G. The use of pressure garments on hypertrophic scars. J Tissue Viability. 2002 Jan;12(1):11-5. doi: 10.1016/s0965-206x(02)80004-3. PMID 11887386
- [Result] Ng CL, Lee ST, Wong KL. Pressure garments in the prevention and treatment of keloids. Ann Acad Med Singap. 1983 Apr;12(2 Suppl):430-5. PMID 6625526
- [Result] Kal HB, Veen RE. Biologically effective doses of postoperative radiotherapy in the prevention of keloids. Dose-effect relationship. Strahlenther Onkol. 2005 Nov;181(11):717-23. doi: 10.1007/s00066-005-1407-6. PMID 16254707
- [Result] Narkwong L, Thirakhupt P. Postoperative radiotherapy with high dose rate iridium 192 mould for prevention of earlobe keloids. J Med Assoc Thai. 2006 Apr;89(4):428-33. PMID 16696385
- [Result] Gusak VK, Fistal' EIa, Speranskii II, Zagoruiko NN. [Cryotherapy of postburn hypertrophic scars]. Klin Khir (1962). 1994;(1-2):15-7. Russian. PMID 8078236
- [Result] Har-Shai Y, Amar M, Sabo E. Intralesional cryotherapy for enhancing the involution of hypertrophic scars and keloids. Plast Reconstr Surg. 2003 May;111(6):1841-52. doi: 10.1097/01.PRS.0000056868.42679.05. PMID 12711943
- [Result] O'Brien L, Pandit A. Silicon gel sheeting for preventing and treating hypertrophic and keloid scars. Cochrane Database Syst Rev. 2006 Jan 25;(1):CD003826. doi: 10.1002/14651858.CD003826.pub2. PMID 16437463
- [Result] Tredget EE, Nedelec B, Scott PG, Ghahary A. Hypertrophic scars, keloids, and contractures. The cellular and molecular basis for therapy. Surg Clin North Am. 1997 Jun;77(3):701-30. doi: 10.1016/s0039-6109(05)70576-4. PMID 9194888